CLINICAL TRIAL: NCT06204848
Title: Acquisition of Imaging Data of Vitreous Opacities in Human Eyes Using a Non-Invasive Imaging Device
Brief Title: Imaging of Vitreous Opacities in a Canadian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PulseMedica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SVO-IDFIH002
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Floaters; Vitreous Opacities
MeSH Terms: conditions — vitreous floaters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imaging using the SVO-ID (Experimental): Patients will have their eyes imaged with the SVO-ID as part of a study visit.
  Interventions: Device: SVO-ID

INTERVENTIONS:
Device: SVO-ID — Combined scanning laser ophthalmoscope (SLO) and optical coherence tomography (OCT) for imaging of the eye

SUMMARY:
The goal of this clinical trial is to capture imaging data of eye floaters in the population to build an imaging database to learn more about them in. Participants will imaged with an investigational ophthalmic imaging device to capture images of their floaters.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Symptomatic vitreous opacities (floaters) in vision
* Clear ocular media, to allow a clear view of the vitreous for the SVO-ID

Exclusion Criteria:

* Younger than 18 years of age
* Presence of vitreous hemorrhage
* Cataract Grade 3 and above
* Opacification of lens, cornea, or vitreous
* Diagnosis of narrow angle glaucoma
* Refractive error is outside the range of -6D to+3D
* Astigmatism is outside the range of +/-2D of cylinder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Successful capture of SLO and OCT imaging data of SVOs for algorithm development | Through study completion, an average of 6-8 months
  Successful collection of SLO and OCT imaging data

SECONDARY OUTCOMES:
Collection of patient-reported symptoms | Through study completion, an average of 6-8 months
  Patient feedback regarding symptoms related to SVOs being imaged

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Retina Consultants, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No